CLINICAL TRIAL: NCT01774019
Title: Randomized Multi-Center Study Comparing No Drainage to Preoperative Biliary Drainage Using Metal Stents in Patients With Resectable Pancreatic or Periampullary Cancer
Brief Title: Preoperative Biliary Drainage in Resectable Pancreatic or Periampullary Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90914721; E7059 (Other: Boston Scientific)
Record Dates: First submitted 2012-10-02; First posted 2013-01-23 (Estimated); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Pancreatic Carcinoma
Keywords: Pancreatic; Periampullary Cancer; Preoperative Biliary Drainage; Resectable
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WallFlex™ Biliary RX Fully Covered/Uncovered Stent System (Active Comparator): Patients in this group will receive a fully covered or uncovered study SEMS (self-expanding metal stent)
  Interventions: Device: WallFlex™ Biliary RX Fully Covered/Uncovered Stent System
- None (No Pre-Operative Biliary Drainage) (No Intervention): Patients in this group will not receive pre-operative biliary drainage with a study SEMS

INTERVENTIONS:
Device: WallFlex™ Biliary RX Fully Covered/Uncovered Stent System
  Arms: WallFlex™ Biliary RX Fully Covered/Uncovered Stent System

SUMMARY:
The purpose of this study is to demonstrate that preoperative biliary drainage using self-expanding metal stents (SEMS) does not negatively impact overall surgical outcomes in patients undergoing pancreaticoduodenectomy for treatment of pancreatic or periampullary cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study
* Diagnosis of probable pancreatic cancer, distal common bile duct (CBD) cholangiocarcinoma and other periampullary cancers (histology not required)
* Biliary obstructive symptoms or signs
* Bilirubin level at/above 100 umol per liter (5.8 mg/dL)
* Distal biliary obstruction consistent with pancreatic cancer, distal CBD cholangiocarcinoma or other periampullary malignancy
* Location of distal biliary obstruction is such that it would allow the proximal end of a stent to be positioned at least 2cm from the hilum
* Patients deemed as resectable by pancreatic protocol CT or MRI
* Surgical candidate per pancreatobiliary surgeon after multi-disciplinary discussion
* Surgery intent within 4 weeks
* Endoscopic and surgical treatment to be provided by same team

Exclusion Criteria:

* Biliary strictures caused by confirmed benign tumors
* Biliary strictures caused by malignancies other than pancreatic cancer, distal CBD cholangiocarcinoma and other periampullary cancers
* Surgically altered biliary tract anatomy, not including prior cholecystectomy
* Neoadjuvant chemotherapy for current malignancy
* Palliative indication due to reasons other than surgical candidate status
* Previous biliary drainage by ERCP/PTC
* Patients for whom endoscopic techniques are contraindicated
* Participation in another investigational trial within 90 days
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Costamagna, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (11):
- Standford University Medical Center, Stanford, California, United States
- Westmead Hospital, Westmead, New South Wales, Australia
- ULB Erasme Hospital, Brussels, Belgium
- China (2):
  - Beijing Friendship Hospital, Beijing
  - Xijing Hospital of Digestive Diseases Fourth Military Medical University, Xi'an
- Hopital Edouard Herriot, Lyon, France
- Hong Kong (2):
  - Queen Elizabeth Hospital, Kowloon
  - Prince of Wales Hospital, the Chinese University of Hong Kong, Shatin
- Asian Institute of Gastroenterology, Hyderabad, India
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy
- Tokyo Medical University, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were screened by site investigators at 11 academic medical centers globally between February 2013 and August 2021.
  The first participant was enrolled in February 2013 and the last participant was enrolled in August 2021.
Pre-assignment Details: Of the 765 participants assessed for eligibility, 284 met criteria and were randomized.
Groups:
- WallFlex™ Biliary RX Fully Covered/Uncovered Stent System: Patients in this group will receive a fully covered or uncovered study SEMS (self-expanding metal stent)
  WallFlex™ Biliary RX Fully Covered/Uncovered Stent System
Period: Overall Study
Arm/Group | WallFlex™ Biliary RX Fully Covered/Uncovered Stent System | None (No Pre-Operative Biliary Drainage)
Started | 144 | 140
Completed | 138 | 136
Not Completed | 6 | 4
Not completed — No longer meets protocol criteria | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Surgery delayed > 120 days | 1 | 0
Not completed — Patient refused surgery | 1 | 1
Not completed — Unable to implant study device | 1 | 0
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WallFlex™ Biliary RX Fully Covered/Uncovered Stent System | None (No Pre-Operative Biliary Drainage) | Total
Number analyzed (Participants) | 144 | 140 | 284
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (11.5) | 64.9 (11.7) | 63.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 59 | 123
  Male | 80 | 81 | 161
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 52 | 51 | 103
  Belgium | 8 | 7 | 15
  United States | 4 | 3 | 7
  Japan | 9 | 7 | 16
  China | 2 | 2 | 4
  Italy | 27 | 27 | 54
  Australia | 3 | 3 | 6
  France | 3 | 3 | 6
  India | 36 | 37 | 73
Height [Mean (Standard Deviation); unit: cm] | 163.3 (9.1) | 161.8 (8.7) | 162.5 (8.9)
Weight [Mean (Standard Deviation); unit: kg] | 65.0 (12.8) | 63.2 (12.7) | 64.1 (12.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (3.9) | 24.1 (3.9) | 24.2 (3.9)
Karnofsky Score (overall health status) [Mean (Standard Deviation); unit: units on a scale] — 100 Normal no complaints nor evidence of disease;90 Normal activity, minor signs/symptoms of disease;80 Normal activity w/effort, some sign/symptom of disease;70 Cares for self, unable to carry on normal activity/do active work;60 Requires occasional assistance, able to care for most personal needs;50 Requires considerable assistance & frequent medical care;40 Disabled, requires special care/assistance;30 Severely disabled, hospitalization indicated, death not imminent;20 Very sick, hospitalization & active support treatment necessary;10 Moribund, fatal processes progress rapidly;0 Dead
  units on a scale | 91.3 (7.3) | 89.6 (9.1) | 90.5 (8.2)
Total serum bilirubin [Mean (Standard Deviation); unit: mg/dl] | 14.0 (6.3) | 12.9 (5.0) | 13.4 (5.7)
Tumor location on imaging Head [Count of Participants; unit: Participants] | 102 | 85 | 187
Tumor location on imaging Ampullary [Count of Participants; unit: Participants] | 30 | 34 | 64
Tumor location on imaging distal [Count of Participants; unit: Participants] | 12 | 16 | 28
Tumor location on imaging Uncinate process [Count of Participants; unit: Participants] | 0 | 2 | 2
Tumor location on imaging Isthmus [Count of Participants; unit: Participants] | 0 | 1 | 1
Tumor location on imaging tail [Count of Participants; unit: Participants] | 0 | 1 | 1
Tumor location on imaging Duodenum [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Pre-operative, Operative and Post-operative Adverse Events to 120 Days Post Randomization or to 30 Days Post Surgery, Whichever Comes Last
Description: The primary end point was all serious adverse events (SAEs), including all preoperative, operative and postoperative adverse events reported from the time of randomization to 120 days post-randomization or 30 days post-CIS (up to 150 days post-randomization), whichever occurred later.
Time Frame: 120 to 150 days
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex™ Biliary RX Fully Covered/Uncovered Stent System | None (No Pre-Operative Biliary Drainage)
Number analyzed (Participants) | 138 | 136
Participants | 40 | 36

2. Secondary Outcome: Stent Placement Success
Description: Stent placement success: ability to deploy the stent in satisfactory position across the stricture (For patients who are randomized to biliary drainage with a metal stent)
Time Frame: Procedure
Population: 3 patients in the WallFlex Biliary RX Fully Covered/Uncovered Stent arm had no stent placed. Patients in the no drainage arm are not intended to have a stent placement per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex™ Biliary RX Fully Covered/Uncovered Stent System | None (No Pre-Operative Biliary Drainage)
Number analyzed (Participants) | 141 | 0
Participants | 140 |

3. Secondary Outcome: Number of Patients With Biliary Re-interventions
Description: Count of patients with biliary interventions after baseline
Time Frame: 120 to 150 days
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex™ Biliary RX Fully Covered/Uncovered Stent System | None (No Pre-Operative Biliary Drainage)
Number analyzed (Participants) | 144 | 140
Participants | 8 | 12

4. Secondary Outcome: Success Rate of Curative Intent Surgery
Description: This is the number of patients that had successful resection
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex™ Biliary RX Fully Covered/Uncovered Stent System | None (No Pre-Operative Biliary Drainage)
Number analyzed (Participants) | 118 | 129
Participants | 103 | 115

5. Secondary Outcome: All-cause Mortality
Description: Mortality which occurs within 150 days of baseline
Time Frame: 150 days
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex™ Biliary RX Fully Covered/Uncovered Stent System | None (No Pre-Operative Biliary Drainage)
Number analyzed (Participants) | 144 | 140
Participants | 11 | 11

ADVERSE EVENTS:
Time Frame: All serious adverse events (SAEs), including all preoperative, operative and postoperative adverse events reported from the time of randomization to 120 days post-randomization or 30 days post-CIS (up to 150 days post-randomization), whichever occurred later.
Arm/Group | WallFlex™ Biliary RX Fully Covered/Uncovered Stent System | None (No Pre-Operative Biliary Drainage)
All-Cause Mortality (participants affected / at risk) | 11/144 | 11/140
Serious Adverse Events (participants affected / at risk) | 40/144 | 36/140
Other Adverse Events (participants affected / at risk) | 0/144 | 0/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WallFlex™ Biliary RX Fully Covered/Uncovered Stent System (N=144) | None (No Pre-Operative Biliary Drainage) (N=140)
Cholangitis (Hepatobiliary disorders) | 4 | 6
Pancreatitis (Gastrointestinal disorders) | 7 | 0
Hemorrhage after ERCP (Vascular disorders) | 3 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 1
Biliary obstruction (Investigations) | 0 | 1
Fever (General disorders) | 4 | 0
Infection (Infections and infestations) | 1 | 0
Left leg swelling (General disorders) | 1 | 0
Persistent jaundice (Hepatobiliary disorders) | 1 | 0
Respiratory infection (Infections and infestations) | 1 | 0
Septic arthritis (Infections and infestations) | 1 | 0
Stroke (Nervous system disorders) | 1 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0
Hemorrhage after CIS (Injury, poisoning and procedural complications) | 3 | 10
Intra-abdominal abscess (Infections and infestations) | 4 | 8
Pancreaticojejunostomy leakage (Injury, poisoning and procedural complications) | 4 | 4
Sepsis (Infections and infestations) | 2 | 4
Biliary leakage (Injury, poisoning and procedural complications) | 2 | 2
Delayed gastric emptying (Gastrointestinal disorders) | 2 | 2
Wound infection (Infections and infestations) | 2 | 2
Ascites (Gastrointestinal disorders) | 1 | 1
Diabetes (Metabolism and nutrition disorders) | 0 | 2
Gastrojejunostomy or duodenojejunostomy leakage (Injury, poisoning and procedural complications) | 0 | 2
Small bowel obstruction (Gastrointestinal disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hemorrhage after ERCP (Vascular disorders) | 1 | 0
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolemia (Vascular disorders) | 1 | 0
Pain (Gastrointestinal disorders) | 0 | 1
Pancreaticogastrostomy leakage (Injury, poisoning and procedural complications) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Refractory shock (Vascular disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Right hemiplegia (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-10-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT01774019/Prot_000.pdf
  • Statistical Analysis Plan (2012-07-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT01774019/SAP_001.pdf